CLINICAL TRIAL: NCT03641794
Title: A Phase I Study of DN1406131 in Healthy Adults
Brief Title: Indoleamine 2,3-Dioxygenase (IDO) Inhibitor in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Collaborators: Shanghai De Novo Pharmatech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DN-DN1406131-101
Record Dates: First submitted 2018-08-15; First posted 2018-08-22 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2018-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DN1406131 (Experimental): 25 mg,50 mg,100 mg,200 mg,400 mg,600 mg,800 mg
  Interventions: Drug: DN1406131
- Placebo (Placebo Comparator): 25 mg,50 mg,100 mg,200 mg,400 mg,600 mg,800 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DN1406131 — IDO1 and TDO2 inhibitor
  Arms: DN1406131
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double blind Phase I study to evaluate the safety, tolerability, and pharmacokinetics of escalating oral doses of DN1406131, an investigational agent intended to inhibit the indoleamine 2,3-dioxygenase 1 (IDO1) enzyme and tryptophan 2,3-Dioxygenase 2 (TDO-2) and help the human immune system attack solid tumor cells more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Age greater of 18 years and less than 45
* Weight ≥50 kg,body mass index of 19~26 kg/m2
* Signed ICF

Exclusion Criteria:

* active autoimmune disease
* uncontrolled concurrent illness
* Smoking
* Drugs
* positive serology for HIV, Hepatitis B or C,Syphilis
* Pregnancy or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
adverse events - type, incidence, severity | 28 day
  Evaluate the safety and toxicity of DN1406131 in healthy volunteers
Maximum Tolerated Dose | 14 day
  To define the Maximum Tolerated Dose (MTD)

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 48 hours
  Cmax
Serum for biomarkers of IDO activity (kynurenine and tryptophan) | 48 hours
  Evaluation of serum for biomarkers of IDO activity (kynurenine and tryptophan), before and after initiation of therapy.
  Pharmacodynamics（PD）
Elimination half-life | 48 hours
  T1/2
peak time | 48 hours
  Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Qinghong Zhou, Study Director — Jiangxi Qingfeng Pharmaceutical Co. Ltd.
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shandong, China